CLINICAL TRIAL: NCT05716399
Title: Effect of Transcutaneous Electrical Stimulation of Acupoints on the Incidence of Hypotension After Spinal Anesthesia in Elderly Patients Undergoing Orthopaedic Surgery
Brief Title: Effect of Acupoint Electrical Stimulation on Incidence of Hypotension After Spinal Anesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Tongji Hospital, Tongji University School of Medicine (Other)
Collaborators: ShuGuang Hospital (Other)
Responsible Party: Principal Investigator, Shaorui Gu, Doctor, Shanghai Tongji Hospital, Tongji University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-984-59-01
Record Dates: First submitted 2023-01-05; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Anesthesia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: In order to ensure the objectivity and reliability of the study, the statistical analysts are blinded, and the subjects and operators are not blind. The operator is responsible for the implementation of anesthesia, the connection and use of TEAS, and data collection; The statistical analyst is responsible for data entry, data sorting and statistical analysis.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Transcutaneous electric stimulation pretreatment group (Experimental): 30 minutes before the implementation of spinal anesthesia, TEAS (density wave 10/50Hz, one side of Neiguan and Quchi points connected to two electrodes on the same wire on the electroacupuncture instrument) was continuously performed on both sides of Neiguan and Quchi points.
  Interventions: Device: Transcutaneous electric stimulation pretreatment
- Transcutaneous acupoint electrical stimulation treatment group (Active Comparator): Within 30 minutes after the occurrence of hypotension, TEAS (density wave 10/50Hz, one side of Neiguan point and Quchi point connected to two electrodes on the same wire on the electroacupuncture instrument) was continuously performed on both sides of Neiguan and Quchi points.
  Interventions: Device: Transcutaneous acupoint electrical stimulation treatment
- Transcutaneous acupoint pseudo electric stimulation group (Sham Comparator): Paste the electrode, turn on the power, but no current output.
  Interventions: Device: Transcutaneous acupoint pseudo electric stimulation

INTERVENTIONS:
Device: Transcutaneous electric stimulation pretreatment — Within 30 minutes before spinal anesthesia or 30 minutes after hypotension, TEAS (density wave 10/50Hz, one side of Neiguan and Quchi points connected to two electrodes on the same wire on the electroacupuncture instrument) was continuously performed on both sides of Neiguan and Quchi points, and the current intensity was only as high as the patient could comfortably tolerate (the electrical stimulation intensity was 2-3 times of the sensory threshold, for example, if the electrical stimulation intensity was 5 mA, 10-15 mA was used for stimulation), Record the specific value of current. FTEAS group pastes electrode piece, turns on the power, but there is no current output.
  Arms: Transcutaneous electric stimulation pretreatment group
Device: Transcutaneous acupoint electrical stimulation treatment — Transcutaneous acupoint electrical stimulation treatment
  Arms: Transcutaneous acupoint electrical stimulation treatment group
Device: Transcutaneous acupoint pseudo electric stimulation — Transcutaneous acupoint pseudo electric stimulation
  Arms: Transcutaneous acupoint pseudo electric stimulation group

SUMMARY:
This study is intended to include elderly patients who are selected to undergo lower limb and pelvic orthopedic surgery under spinal anesthesia. Through prospective, randomized and controlled clinical trials, the investigators will observe the effect of this treatment on the incidence of hypotension in elderly patients after spinal anesthesia through TEAS points Neiguan and Quchi before or during surgery, and further explore its related mechanisms.

DETAILED DESCRIPTION:
Research content: This study aims to observe whether TEAS intervention on Neiguan (PC-6) and Quchi (LI-11) before and during operation can improve the incidence and degree of hypotension after spinal anesthesia, as well as the changes of neurotransmitters and related hormones in blood.

Research methods:

* 111 elderly patients (including hip or lower limb fractures, hip and knee joint replacement or debridement) who were selected for lower limb or pelvic surgery under spinal anesthesia were randomly divided into percutaneous point electrical stimulation pretreatment group (PTEAS group), percutaneous point electrical stimulation treatment group (TEAS group) and percutaneous point pseudo electrical stimulation group (FTEAS group).

  * After entering the operating room, the vital signs were monitored routinely, and the volume was evaluated by measuring the variability of the inferior vena cava with ultrasound before anesthesia. Then, the radial artery was punctured and catheterized, and sodium lactate was infused (8ml/Kg).

    * Within 30 minutes before spinal anesthesia or 30 minutes after hypotension, TEAS (density wave 10/50Hz, one side of Neiguan and Quchi points connected to two electrodes on the same wire on the electroacupuncture instrument) was continuously performed on both sides of Neiguan and Quchi points, and the current intensity was only as high as the patient could comfortably tolerate (the electrical stimulation intensity was 2-3 times of the sensory threshold, for example, if the electrical stimulation intensity was 5 mA, 10-15 mA was used for stimulation), Record the specific value of current. FTEAS group pastes electrode piece, turns on the power, but there is no current output.

      * Select L2/3 or L3/4 interval for spinal anesthesia, use 0.75% cloth ratio, and the dose standard is 0.025ml/Kg.

        * Collect venous blood after entering the operating room and 30 minutes after anesthesia to measure the levels of neurotransmitters and hormones, record the baseline value of vital signs and changes during operation, observe the occurrence and treatment of adverse events during operation, and follow up the troponin T level and the incidence of delirium after operation.

          * Remedial measures for clinical safety:

When severe hypotension occurs during operation, which leads to irreversible adverse effects, it needs to be intervened by multiple means.

Those who are diagnosed as delirium through CAM determination shall be treated with haloperidol or dexmedetomidine.

ELIGIBILITY:
Inclusion Criteria:

* 90>65, regardless of gender;

  * ASA classification I-III; ③ Orthopedic surgery was performed under spinal anesthesia; ④ Sign the informed consent form.

Exclusion Criteria:

* Uncontrolled hypertension;

  * Arrhythmia or myocardial ischemia;

    * Severe cardiopulmonary insufficiency;

      * HB<100g/L;

        * Severe dehydration; ⑥ There are contraindications to spinal anesthesia; ⑦ Allergies to local anesthetics;

          * Communication barriers; ⑨ Refusing to sign the informed consent form.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 111 (Estimated)
Dates: Start 2023-02-20 (Estimated); Primary Completion 2023-12-20 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of hypotension | 30 mins after anesthesia
  30 mins after anesthesia, hypotension was defined as MAP<25% of the baseline value

CONTACTS AND LOCATIONS:
Overall Officials: Wenli Wang, Doctor, Principal Investigator — Shanghai Tongji Hospital, Tongji University School of Medicine

IPD SHARING:
Plan to Share IPD: No